CLINICAL TRIAL: NCT06367920
Title: Multicenter Study on Rehabilitation Medical Data for Pediatric Big Brain
Brief Title: Multicenter Study on Rehabilitation Medical Data for Pediatric Big Brain Development
Status: Recruiting | Type: Observational
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Principle investigator, Bundang CHA Hospital
Other Study IDs: 2022-02-005
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Pediatric ALL; Healthy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging, Behavioral assessments — Magnetic Resonance Imaging, Behavioral assessments

SUMMARY:
Retrospective study for development of imaging-genetics (brain imaging/genome big data) models and algorithms that are clinically explainable and have high predictive performance in brain research on pediatric developmental disorders

DETAILED DESCRIPTION:
Retrospective study for development of imaging-genetics (brain imaging/genome big data) models and algorithms that are clinically explainable and have high predictive performance in brain research on pediatric developmental disorders

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects and patients 20 years old or younger who underwent imaging examinations performed at the Department of Rehabilitation Medicine at our hospital from January 2010 to December 2023 (patients who underwent brain MRI tests to determine the cause of developmental delay)

Exclusion Criteria:

* None

Max Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy subjects and patients 20 years old or younger who underwent imaging examinations performed at the Department of Rehabilitation Medicine at our hospital from January 2010 to December 2023 (patients who underwent brain MRI tests to determine the cause of developmental delay)
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain magnetic resonance imaging | A time point at which imaging was performed between January 1, 2010 and December 31, 2024
  MRI scan is a process of measuring anatomical changes of brain and tract fiber

SECONDARY OUTCOMES:
Medical records | A time point at which recording medical examinations was performed between January 1, 2010 and December 31, 2024
  Medical records including basic characteristics and behavioral assessments

CONTACTS AND LOCATIONS:
Overall Officials: Minyoung Kim, M.D., Ph.D., Principal Investigator — Bundang CHA Hospital
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea